CLINICAL TRIAL: NCT04788342
Title: Pulse Wave Parameters Registered by a Single-lead Electrocardiogram Monitor With Photoplethysmography Function in the Assessment of Systolic Function of the Left Ventricle.
Brief Title: Pulse Wave Parameters in the Assessment of Systolic Function of the Left Ventricle.
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: S17022021
Record Dates: First submitted 2021-02-16; First posted 2021-03-09 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-02

CONDITIONS: Hypertension; Heart Failure
Keywords: pulse wave; systolic function of the left ventricle; ejection fraction; blood pressure; a single-lead electrocardiogram; remote determination of the systolic function
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — Echocardiography; Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with and without left ventricular systolic dysfunction: Patients with different pathologies of the cardiovascular system (coronary artery disease, hypertension, valvular heart disease, heart failure) will be performed pulse wave recording using a CardioQvark cardiomonitor and echocardiography.
  Interventions: Device: pulse wave recording, echocardiography.

INTERVENTIONS:
Device: pulse wave recording, echocardiography. — pulse wave recording using a single-channel electrocardiogram cardiomonitor with photoplethysmography, conducting echocardiography according to a standard protocol with the determination of systolic function of the left ventricle
  Other Names: blood pressure measurement

SUMMARY:
This is a prospective, single-center, non-randomized, observational study. The aim of this study is to determine the potential of a single-lead electrocardiogram monitor CardioQvark with photoplethysmography function use to evaluate systolic function of the left ventricle.

The study is conducted in the clinic of I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia. It is planned to include 400 patients. Recording of the electrocardiogram and photoplethysmogram by the monitor CardioQvark and the assessment of systolic function using echocardiography will be performed in all study participants.

The result of this study will be the identification of the parameters of the pulse wave and electrocardiogram that will correlate with systolic function of the left ventricle. It is also planned to determine the diagnostic effectiveness of this method.

DETAILED DESCRIPTION:
The aim of this study is to determine the potential of a single-lead electrocardiogram (ECG) monitor CardioQvark (Moscow, Russia) with photoplethysmography function use to evaluate parameters systolic function of the left ventricle. Also according to the photoplethysmogram (PPG), using a special algorithm, the levels of systolic and diastolic blood pressure are calculated.

The single-lead electrocardiogram monitor CardioQvark (it is registered with the Federal Service for Health Supervision on February 15, 2019. RZN (Roszdravnadzor) No. 2019/8124) looks like an iPhone cover and records electrocardiogram (I standard lead) and photoplethysmogram (pulse wave) simultaneously.

This is a prospective, single-center, non-randomized, observational study. The investigators are planning to include in the study 400 patients with different pathologies of the cardiovascular system (coronary artery disease, hypertension, valvular heart disease, heart failure) according to the inclusion criteria.

Collection of medical history; physical examination (including inspection, palpation and auscultation, as well as determination of breathing rate, pulse rate, height, and weight) will be performed for the entire group of patients. Electrocardiogram and photoplethysmogram registration and assessment of the blood pressure using a CardioQvark monitor will be performed on all study participants at rest (the patient will sit quietly for 10-15 minutes before the examination). The reference blood pressure will be measured using a cuff-based blood pressure device ("Microlife BP AG1-10") that is worn on the upper arm according to the World Health Organization recommendations.

All subjects will undergo an echocardiography ("Dimension/Vivid 7 PRO General Electric Medical System"), the examination will be performed by an experienced doctor (the doctor will not have data on the parameters of the pulse wave and electrocardiogram). The extended protocol echocardiography will be performed according to the recommendations of European Association of Cardiovascular Imaging (EACVI) and American Society of Echocardiography (ASE). All examinations will be performed consistently within one day.

All electrocardiograms and photoplethysmograms records will be sent to the CardioQVARK server and processed by the algorithm using signal processing based on the wavelet transformation. Then engineers of "CardioQvark" (Limited Liability Company) will calculate the pulse wave parameters:

* B1 is the beginning of the wave
* B0 is the point of maximum increase of the anterior front
* SEP is the peak of the ejected pulse wave
* DER3 is the first positive peak of the third derivative
* SEPMAX is the point of the first inflection of pulse wave
* SRP is the peak of the reflected systolic wave
* DP is the peak of the diastolic wave
* End is the end of the wave
* perfusion index
* augmentation index.

A spectral analysis of the electrocardiogram will be performed using a continuous wavelet transform, the principles of which are based on the Fourier transform:

* TpTe - time from peak to end of the T-wave
* VAT - time from the beginning of the QRS to the R-peak
* QTc - corrected QT interval.
* QT / TQ - the ratio of QT length to TQ length (from the end of T to the beginning of the QRS of the next complex).
* QRS_E - the total energy of the QRS wave based on the wavelet transform
* T_E - T-wave total energy based on wavelet transform
* TP_E- energy of the main tooth of the T-wave based on the wavelet transform
* BETA, BETA_S - T-wave asymmetry coefficients (simple and smooth versions)
* BAD_T - flag of T-wave quality (whether expressed in the current lead
* QRS_D1_ons - energy of the leading edge of the R-wave (based on the "first derivative" wavelet transform)
* QRS_D1_offs - energy of the trailing edge of the R-wave (based on the "first derivative" wavelet transform)
* QRS_D2 - peak energy of the R-wave (based on the "second derivative" wavelet transform)
* QRS_Ei (i = 1,2,3,4) - QRS-wave energy in 4 frequency ranges (2-4-8-16-32 Hz) based on wavelet transform
* T_Ei (i = 1,2,3,4) - T-wave energy in 4 frequency ranges (2-4-6-8-10 Hz) based on wavelet transform
* HFQRS - the amplitude of the RF components of the QRS wave. The engineers will not have echocardiography results.

The investigators will evaluate parameters of the pulse wave (photoplethysmogram) and electrocardiogram and compare the results with echocardiography (ejection fraction, left ventricular outflow tract velocity time integral (VTI), left ventricular global longitudinal strain (GLS)).The mathematical model for determining the systolic dysfunction of the left ventricle will be built on the basis of the parameters of the photoplethysmogram and the electrocardiogram.

Intergroup analysis of significant differences, correlation analysis and Bland-Altman method will be used for statistical data analysis. All statistical analyses will be perform using a computer program for statistical processing of data SPPS (statistical package for the social sciences) Statistics Version 26.

It is planned to obtain comparative characteristics of the pulse wave and electrocardiogram parameters registered by the CardioQvark monitor and the indicators of systolic function of the left ventricle detected during echocardiography. The result of this study will be the identification of the parameters of the pulse wave and electrocardiogram that will correlate with systolic dysfunction of the left ventricle. It is planned to determine the diagnostic effectiveness of this method. The accuracy of the blood pressure measurement using the CardioQvark monitor will also be evaluated.

Thus, a quick and convenient assessment of systolic function of the left ventricle and blood pressure measurement will be available. So, study results will improve the diagnosis and treatment of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of written informed consent of the patient to participate in the study.
2. The presence of diagnosed cardiac pathology according anamnesis (coronary artery disease (I-IV classes according Canadian Cardiovascular Society grading of angina pectoris, post myocardial infarction, patients after percutaneous coronary intervention or coronary artery bypass grafting); hypertension (stages I- III); valvular heart disease (except patients with aortic valve stenosis and mechanical prosthetic heart valve); heart failure (I-IV NYHA).

   -

   Exclusion Criteria:

1. Patient's reluctance to participate in the study. 2. Poor quality of ECG recording by a single-channel ECG monitor. 3. Poor visualization of the heart during echocardiography.

-

Non-inclusion criteria:

1. The presence of rhythm and conduction disorders (WPW syndrome, frequent premature ventricular complexes, 2nd and 3rd degree sinoatrial block, 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block).
2. Patients with permanent cardiac pacemaker, cardio-resynchronization therapy (CRT), implantable cardioverter-defibrillator (ICD).
3. Conditions that can impair ECG recording quality (Parkinson's disease, essential tremor, etc.) or conditions that make it difficult to record ECG and photoplethysmogram (traumatic arm amputation)
4. Mental illness (diagnosed early)
5. Diseases with a life expected expectancy of less than 2 years.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with different pathologies of the cardiovascular system (coronary artery disease, hypertension, valvular heart disease, heart failure) aged 18 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Determination of the comparative characteristics of the pulse wave parameters registered by a single- lead ECG monitor CardioQvark and indicators of systolic function of the left ventricle detected during echocardiography. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Diagnostic accuracy of the pulse wave and electrocardiogram parameters registered by a single- lead ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Determination of the sensitivity of left ventricular systolic dysfunction detected by analysis of the pulse wave and electrocardiogram registered by a single- lead ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Determination of specificity of left ventricular systolic dysfunction detected by analysis of the pulse wave and electrocardiogram registered by a single- lead ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Determination of prognostic value of positive and negative results of left ventricular systolic dysfunction detected by analysis of the pulse wave and electrocardiogram registered by a single-channel ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Determination of area under receiver operating characteristic curve of left ventricular systolic dysfunction detected by analysis of the pulse wave and electrocardiogram registered by a single- lead ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
Determination of correlation coefficient of left ventricular systolic dysfunction detected by analysis of the pulse wave and electrocardiogram registered by a single-channel ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of left ventricular systolic dysfunction detected by echocardiography with the results of the presence of left ventricular systolic dysfunction obtained using the mathematical model of pulse wave and electrocardiogram parameters.
assessment of the accuracy of the blood pressure measurement using a single-channel ECG monitor CardioQvark. | Through study completion, an average of 1 year.
  comparison of blood pressure values obtained on the basis of a mathematical model of pulse wave parameters and measured using a cuff-based device.

SECONDARY OUTCOMES:
significance of the parameter TpTe on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter VAT on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QTc on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QT / TQ on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_E on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter T_E on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter TP_E on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BETA on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BETA_S on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter BAD_T on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D1_ons on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D1_offs on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_D2 on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter QRS_Ei on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter T_Ei on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter HFQRS on the ECG in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  an ECG spectral analysis will be performed using the Fourier Transform
significance of the parameter B1 on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter B0 on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter SEP on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter DER3 on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter SEPMAX on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter SRP on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter DP on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark
significance of the parameter perfusion index on the pulse wave in the determination of left ventricular systolic dysfunction | Through study completion, an average of 1 year.
  the analysis of the pulse wave registered by a single-lead ECG monitor with the photoplethysmography CardioQvark

CONTACTS AND LOCATIONS:
Overall Officials: Petr Chomakhidze, Professor, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University); Zhanna Sagirova, Graduate, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The research sponsor is Sechenov University. Data disclosure is not permitted by the local ethics committee. For more information about the study, you need to contact the principal investigator.